CLINICAL TRIAL: NCT01070147
Title: A Computerized Asthma Management System in the Pediatric Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 100189
Record Dates: First submitted 2010-02-10; First posted 2010-02-17 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Asthma
Keywords: asthma; emergency medicine; medical informatics; computerized reminder systems
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Control (Experimental): The control group will receive a paper-based printed asthma guideline.
  Interventions: Other: Computerized Asthma Management System

INTERVENTIONS:
Other: Computerized Asthma Management System — The intervention group's clinicians will receive prompts via the computerized management system to prompt them for scoring, assessments, and disposition decisions.

SUMMARY:
The primary goal of this study is that the combination of a computerized asthma reminder system with implementation of an guideline will increase utilization and adherence of guideline-driven care, leading to improved patient outcomes.

Hypothesis: An automatic, computerized reminder system for detecting asthma patients in the pediatric ED will increase guideline adherence compared to paper-based guideline.

The specific aims of the study are:

Aim 1: Develop, implement, and integrate the asthma guideline in the ED information system infrastructure.

Aim 2: Evaluate the effect of the asthma detection system combined with the computerized guideline versus the asthma detection system combined with the paper-based guideline.

DETAILED DESCRIPTION:
Asthma is the leading chronic childhood disease affecting 9 million children (12.5%) under 18 years of age (1). Asthma exacerbations cause an estimated 14 million missed school days (2) and more than 1.8 million emergency department (ED) visits annually (2), and account for >60% of asthma-related costs (3). The chronic characteristic of asthma carries a considerable economic burden.

Uncontrolled asthma can lead to exacerbations requiring the patient to seek immediate care, frequently in an ED setting. Several asthma guidelines, including the nationally accepted guideline from the National Heart, Lung, and Blood Institute (NHLBI), exist to support clinicians in providing adequate treatment. Utilization of and adherence with asthma guidelines improves patients' clinical care (4, 5). However, guideline adherence remains suboptimal. In the ED, early recognition and accurate assessment of the severity of airway obstruction and response to therapy are fundamental to the improvement of health for patients with asthma. The NHLBI guidelines emphasize early recognition and treatment of asthma exacerbations, as well as appropriate treatment stratified by severity.

Computer applications for patient care can address barriers to optimal medical care. Computer systems have improved the use and adherence to practice guidelines, provide clinical alerts and reminders, and generate patient-specific treatment recommendations and educational material. Implementation of guideline-driven decision support is frequently paper-based or computerized. In either form a major barrier remains on the busy clinicians to remember to initiate the guideline a process and to embed the guideline tasks in the clinical workflow of the care team (5). The proposed study examines the benefits of a novel approach for reminding clinicians in an ED setting to use guideline-driven care. The approach will apply a workflow-embedded process taking advantage of an advanced information technology infrastructure. The informatics approach will include two elements: a) a computerized, real-time reminder system, which will automatically detect guideline-eligible patients without requiring additional data entry, and b) a computerized, workflow-embedded guideline implementation.

ELIGIBILITY:
Inclusion Criteria:

* all patients aged 2-18 years
* Emergency Severity Index 2 to 5
* availability of completed computerized triage documentation.

Exclusion Criteria:

* critically ill patients (Emergency Severity Index 1)
* patients who leave-without-being seen
* patients who leave against-medical-advice
* patients whose final diagnosis was not asthma (false positive identification by the detection system) or were determined not to be eligible for the guideline.

Ages: 2 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1631 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2015-12-07 (Actual); Study Completion 2015-12-07 (Actual)

PRIMARY OUTCOMES:
length of stay | 48 hours (or patient discharged from emergency department)

SECONDARY OUTCOMES:
guideline adherence | during ED visit (48 hours or less)
number of asthma scores | during ED visit (48 hours or less)

CONTACTS AND LOCATIONS:
Overall Officials: Judith W Dexheimer, MS, Study Director — Vanderbilt University; Dominik Aronsky, MD, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt Children's Hospital, Nashville, Tennessee, United States

REFERENCES:
- [Background] Ref: QuickStats: Percentage of Children Aged <18 years Who Have Ever Had Asthma Diagnosed, by Age Group --- United States, 2003; MMWR April 29, 2005 / 54(16);412. http://www.cdc.gov/mmwr/preview/mmwrhtml/mm5416a5.htm
- [Background] Allergy & Asthma Advocate. Quarterly patient newsletter of the American Academy of Allergy, Asthma and immunology. 2004.
- [Background] Grimshaw JM, Eccles MP, Walker AE, Thomas RE. Changing physicians' behavior: what works and thoughts on getting more things to work. J Contin Educ Health Prof. 2002 Fall;22(4):237-43. doi: 10.1002/chp.1340220408. PMID 12613059
- [Background] Guidelines for the diagnosis and management of asthma. National Heart, Lung, and Blood Institute. National Asthma Education Program. Expert Panel Report. J Allergy Clin Immunol. 1991 Sep;88(3 Pt 2):425-534. No abstract available. PMID 1890276
- [Background] Scribano PV, Lerer T, Kennedy D, Cloutier MM. Provider adherence to a clinical practice guideline for acute asthma in a pediatric emergency department. Acad Emerg Med. 2001 Dec;8(12):1147-52. doi: 10.1111/j.1553-2712.2001.tb01131.x. PMID 11733292